CLINICAL TRIAL: NCT01137019
Title: Optical Coherence Tomography Assessment of Intimal Tissue and Malapposition: A Randomized Comparison of the Biolimus A9-eluting and Everolimus-eluting Coronary Stents
Brief Title: Optical Coherence Tomography Assessment of Intimal Tissue and Malapposition
Acronym: OPTIMA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr Peter Barlis (Other)
Collaborators: Biosensors International (Other)
Responsible Party: Sponsor-Investigator, Dr Peter Barlis, Associate Professor of Medicine, Principal Investigator, Northern Hospital, Australia
Organization: Northern Hospital, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPTIMA A19/10
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Heart Disease
Keywords: Drug-eluting stents; Tomography, Optical Coherence
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biolimus-eluting stent (Active Comparator)
  Interventions: Device: Biolimus-eluting stent
- Everolimus-eluting stent (Active Comparator)
  Interventions: Device: Everolimus-eluting coronary stent

INTERVENTIONS:
Device: Biolimus-eluting stent — The biolimus-eluting coronary stent contains a stainless steel platform on which an abluminally coated polylactic acid (PLA) biodegradable polymer is placed that eludes biolimus-A9.
  Other Names: Biomatrix Flex (Biosensors International)
  Arms: Biolimus-eluting stent
Device: Everolimus-eluting coronary stent — The everolimus-eluting coronary stent is a cobalt chromium platform stent with a permanent fluorinated copolymer matrix that eludes everolimus
  Other Names: Promus (BSC)
  Arms: Everolimus-eluting stent

SUMMARY:
The purpose of this study is to use a high-resolution intracoronary imaging modality, called optical coherence tomography (OCT) to examine two different types of coronary artery stents used to treat patients with coronary artery disease.

DETAILED DESCRIPTION:
The development of coronary stents has significantly improved the safety and efficacy of percutaneous coronary intervention (PCI) compared to balloon angioplasty alone. Nevertheless, restenosis is still encountered in 20 to 40% of coronary lesions after implantation of bare metal stents, inferring frequent repeat revascularization procedures with a negative impact on quality of life and health care expenditures. Drug-eluting stents (DES), with their controlled release of therapeutic agents, have significantly reduced the rate of major adverse cardiac events (MACE) following coronary stent implantation, primarily by a reduction in restenosis and target lesion revascularization.

Optical coherence tomography (OCT) is an optical analogue of intravascular ultrasound (IVUS): it uses an infrared light source (wavelength 1310nm) and measures the backscatter of light in a technique similar to conventional ultrasound. With this technique a resolution up to 10μm in-vivo has been reported, a far better level of resolution compared with IVUS. Optical coherence tomography has been used in vivo and has detected early atherosclerotic plaques previously not visualised by IVUS. Segments with strut malapposition and the presence or thickness of neointimal hyperplasia can also be more accurately assessed with OCT compared with IVUS.

The present study will utilize the imaging capabilities of OCT to assess stent strut malapposition and tissue coverage in two different types of DES. The biolimus-eluting stent eludes biolimus from a biodegradable polylactic acid polymer on the abluminal surface of a stainless steel stent. This stent will be compared in a randomized fashion to the permanent polymer based everolimus-eluting coronary stent made of cobalt chromium alloy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, and acute coronary syndromes including non-ST elevation myocardial infarction
* Presence of one or more coronary artery stenosis > 50% in a native coronary artery with a reference diameter ranging from 2.25 to 4.0 mm which can be covered with one or multiple stents
* No limitation to the number of treated lesions, number of vessels or lesion length according to the randomization group

Exclusion Criteria:

* Known intolerance to aspirin, clopidogrel, heparin, stainless steel, cobalt chromium, Biolimus, everolimus, contrast material
* Acute ST-segment elevation myocardial infarction
* Bypass graft
* Inability to provide informed consent
* Pregnancy
* Planned surgery within 12 months of PCI unless dual antiplatelet therapy is maintained throughout the peri-surgical period
* Left ventricular ejection fraction < 25%
* Serum creatinine > 180mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Rate of stent strut malapposition | 0 Days
  Apposition will be examined immediately following stent implantation following angiographic optimization of stent deployment
Rate of stent strut tissue coverage | At follow-up (one of either 3, 6, 12 or 15 months)
  Subjects will be randomized to follow-up at either one of the time points post stenting (3, 6, 12 or 15 months).

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Barlis, MBBS PhD FRACP, Principal Investigator — Northern Hospital, Department of Cardiology, Victoria, Australia
Locations (1):
- The Northern Hospital, Epping, Victoria, Australia

REFERENCES:
- [Background] Barlis P, Regar E, Serruys PW, Dimopoulos K, van der Giessen WJ, van Geuns RJ, Ferrante G, Wandel S, Windecker S, van Es GA, Eerdmans P, Juni P, di Mario C. An optical coherence tomography study of a biodegradable vs. durable polymer-coated limus-eluting stent: a LEADERS trial sub-study. Eur Heart J. 2010 Jan;31(2):165-76. doi: 10.1093/eurheartj/ehp480. Epub 2009 Nov 4. PMID 19889649
- [Background] Barlis P, van Soest G, Serruys PW, Regar E. Intracoronary optical coherence tomography and the evaluation of stents. Expert Rev Med Devices. 2009 Mar;6(2):157-67. doi: 10.1586/17434440.6.2.157. PMID 19298163
- [Background] Barlis P, Dimopoulos K, Tanigawa J, Dzielicka E, Ferrante G, Del Furia F, Di Mario C. Quantitative analysis of intracoronary optical coherence tomography measurements of stent strut apposition and tissue coverage. Int J Cardiol. 2010 May 28;141(2):151-6. doi: 10.1016/j.ijcard.2008.11.204. Epub 2009 Jan 19. PMID 19155076
- [Background] Tanigawa J, Barlis P, Dimopoulos K, Dalby M, Moore P, Di Mario C. The influence of strut thickness and cell design on immediate apposition of drug-eluting stents assessed by optical coherence tomography. Int J Cardiol. 2009 May 15;134(2):180-8. doi: 10.1016/j.ijcard.2008.05.069. Epub 2008 Sep 4. PMID 18775576